CLINICAL TRIAL: NCT01660204
Title: Antibiotic Treatment of Community-acquired Pneumonia: a Prospective Comparison of Dutch Guideline Advices.
Brief Title: Community-Acquired Pneumonia - Study on the Initial Treatment With Antibiotics of Lower Respiratory Tract Infections
Acronym: CAP-START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, MJM Bonten, Professor, UMC Utrecht
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10-148; 80-82310-97-12044 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2012-05-02; First posted 2012-08-08 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Community-acquired Pneumonia
Keywords: pneumonia, anti-bacterial agents, (cost)efficacy
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Betalactam monotherapy (Active Comparator): Preferred empirical treatment for patients in this arm is Beta-lactam monotherapy e.g. co-amoxiclav or ceftriaxone
  Interventions: Other: Preferred empirical treatment
- Betalactam combination with macrolide (Active Comparator): Preferred empirical treatment for patients in this arm is beta-lactam combination therapy with a macrolide e.g. ceftriaxone and erythromycin
  Interventions: Other: Preferred empirical treatment
- Quinolone monotherapy (Active Comparator): Preferred empirical treatment for patients in this arm is quinolone monotherapy e.g. moxifloxacin or levofloxacin
  Interventions: Other: Preferred empirical treatment

INTERVENTIONS:
Other: Preferred empirical treatment — The investigators are using a cluster-randomized cross-over design for preferred empirical treatment. One of the 3 treatment arms is used as preferred empirical therapy during a period of 4 consecutive months, after which preferred treatment will rotate to 1 of the other 2 regimens. The order of change is randomised per hospital, thereby controlling for inter-hospital variables and minimizing seasonal influences.

SUMMARY:
The purpose of this study is to compare the cost(effectiveness) of three existing antibiotic strategies for patients with community-acquired pneumonia admitted to the hospital, but not the ICU.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to one of the participating hospitals needing treatment for CAP, not being admitted to the ICU are eligible for study inclusion.
* Admission is defined as hospital stay for more than 24 hours.

Exclusion Criteria:

* Patients who are readmitted with CAP within 2 weeks after a previous episode are not eligible.
* Patients with cystic fibrosis are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2283 (Actual)
Dates: Start 2011-02; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Day 90 Mortality | 90 days from admission
  We will assess all-cause mortality on day 90 from admission from the municipal personal records database

SECONDARY OUTCOMES:
Length of intravenous antibiotic treatment | Participants will be followed for the duration of hospital stay, an expected average of 1 week
Length of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 1 week
Tolerability | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Side-effects and complications from antibiotic therapy are registered from clinical record
Complications | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Complications of pneumonia during admission are registered from clinical record.
Health care costs and non-health care costs | 28 days from admission
  Health care costs and non-health care costs are assessed using a short questionnaire 28 days from admission

CONTACTS AND LOCATIONS:
Overall Officials: Marc J. Bonten, MD PhD, Principal Investigator — UMC Utrecht
Locations (7):
- Netherlands (7):
  - Medical Center Alkmaar, Alkmaar
  - AMC Amsterdam, Amsterdam
  - Amphia Hospital Breda, Breda
  - Kennemer Gasthuis, Haarlem
  - Spaarne Hospital, Hoofddorp
  - Diakonessenhuis Utrecht, Utrecht
  - UMC Utrecht, Utrecht

REFERENCES:
- [Derived] Postma DF, Spitoni C, van Werkhoven CH, van Elden LJR, Oosterheert JJ, Bonten MJM. Cardiac events after macrolides or fluoroquinolones in patients hospitalized for community-acquired pneumonia: post-hoc analysis of a cluster-randomized trial. BMC Infect Dis. 2019 Jan 7;19(1):17. doi: 10.1186/s12879-018-3630-7. PMID 30612559
- [Derived] van Werkhoven CH, Postma DF, Mangen MJ, Oosterheert JJ, Bonten MJ; CAP-START study group. Cost-effectiveness of antibiotic treatment strategies for community-acquired pneumonia: results from a cluster randomized cross-over trial. BMC Infect Dis. 2017 Jan 10;17(1):52. doi: 10.1186/s12879-016-2179-6. PMID 28068956
- [Derived] Postma DF, van Werkhoven CH, van Elden LJ, Thijsen SF, Hoepelman AI, Kluytmans JA, Boersma WG, Compaijen CJ, van der Wall E, Prins JM, Oosterheert JJ, Bonten MJ; CAP-START Study Group. Antibiotic treatment strategies for community-acquired pneumonia in adults. N Engl J Med. 2015 Apr 2;372(14):1312-23. doi: 10.1056/NEJMoa1406330. PMID 25830421
- [Derived] van Werkhoven CH, Postma DF, Oosterheert JJ, Bonten MJ. Antibiotic treatment of moderate-severe community-acquired pneumonia: design and rationale of a multicentre cluster-randomised cross-over trial. Neth J Med. 2014 Apr;72(3):170-8. PMID 24846935